CLINICAL TRIAL: NCT02457832
Title: Optimizing Motor Training in Parkinson Disease Through Neural Mechanisms (NEURODEGEN)
Brief Title: Motor Training in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N0870-W
Record Dates: First submitted 2015-05-21; First posted 2015-05-29 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Magnetic Resonance Imaging; Neurology; Neurosciences; Physical Medicine; Parkinson Disease; Rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — Behavior Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Internal guidance training (IG) (Experimental): Adapted tango dancing is a sophisticated, yet accessible system of tactile communication that conveys motor intentions and goals between a leader and follower. Those in IG training will choose direction, timing and amplitude of each successive step, and will communicate this information to their partner through moving their frame and center of mass.
  Interventions: Behavioral: Adapted Tango Dancing
- Externally guided training (EG) (Experimental): Those in EG will learn to attend to sensory cues for movement direction, timing and amplitude of steps, communicated from their partner to them via the frame and center of mass. The 'follower' will wait to receive the movement cue before moving.
  Interventions: Behavioral: Adapted Tango Dancing
- Behavioral Control (BC) (Active Comparator): BC participants will attend group health education sessions adapted to the needs of individuals with PD, about pharmacological management, nutrition, sleep disorders, cognitive deficits, bereavement coping, mobility, balance and home safety. Participants in this training will be instructed not to change their habitual exercise routines. After completing health education, participants will be assigned to an IG or EG training class but will not undergo evaluations.
  Interventions: Behavioral: Behavioral Control (BC) Condition
- Normal Control (NC) (No Intervention): Age-matched controls without Parkinson's disease will come in for a single assessment including MRI.

INTERVENTIONS:
Behavioral: Adapted Tango Dancing — Composed of simple steps, tango involves frequent movement initiation and cessation, multi-directional perturbations and varied rhythms. Participants focus on trunk control and stepping strategies, coordination, somatosensory awareness, attention to partner, path of movement, and aesthetics. Sessions will begin with a typical dance class warm-up consisting of breathing, limbering and postural alignment to upbeat music. Novel step elements will be introduced every class period. Those with PD will partner with an individual without PD. After novel step introduction, the instructor will present rhythmic training, which is indispensable to partnered dancing. Participants will learn 'typical' rhythms from tango and Latin dances, based upon the system of quicks (Q) and slows (S), ubiquitously used in ballroom dance training to understand the temporal relationship of movement to music.
  Arms: Externally guided training (EG); Internal guidance training (IG)
Behavioral: Behavioral Control (BC) Condition — Group health education sessions adapted to the needs of individuals with PD, about pharmacological management, nutrition, sleep disorders, cognitive deficits, bereavement coping, mobility, balance and home safety.
  Arms: Behavioral Control (BC)

SUMMARY:
The purpose of this research study is to learn more about brain activity when individuals with and without Parkinson disease (PD) move their lower limbs. The investigators also want to see if and how two different types of partnered dance affect brain activity in individuals with and without PD. Testing will take place at the Atlanta VA Medical Center and at Emory University. The investigators expect to enroll about 140 people for this study over a five-year period.

DETAILED DESCRIPTION:
Persons with Parkinson's disease (PD) have impaired mobility, which adversely affects their quality of life. The effectiveness of adapted tango dance, in which participants both lead (internally guide: IG) and follow (externally guide: EG) movement has been shown. To improve outcomes in those with PD, the underlying brain mechanisms for both motor impairments and improvement must be studied. IG and EG movements have distinct brain activity patterns. Individuals with PD have trouble with IG movement but this problem is helped by strategies used while "leading." During "following", participants with PD can use many external cues, which helps movement in PD, because EG tasks bypass the basal ganglia, the part of the brain affected by PD. In older persons with PD, the investigators aim to:

* determine brain activation patterns during IG and EG foot movement.
* look into effects of IG and EG training on brain activation along with mobility improvements.

The investigators will begin with a functional Magnetic Resonance Imaging test in a scanner. The investigators will look at brain area correlates of a clinically-used foot-tapping task, during IG and EG conditions in older persons with and without PD. Then, the investigators will assess the relative effectiveness of IG versus EG training during an adapted tango class, compared to a group that participates in health education, for improved mobility and foot tapping. Participants with PD will be assessed for disease severity. They will receive tests of outcome measures while "OFF" and "ON" PD-specific medications at the following time points:

* 1 week before training
* 1 week after training
* 1 month after training Participants must attend 20 lessons of IG or EG adapted tango in 12 weeks, taught by an experienced instructor. In the functional MRI (fMRI) scanner, the investigators will assess participants for improved foot tapping after training. The investigators will also look at changes in activation in specific brain circuits along with training effects upon mobility.

The long-term goal is to improve motor training as much as possible for persons with PD by understanding foot movement brain circuitry in PD as well as brain changes in circuitry through which training is effective. This work proposes to illumine information about brain function that is very important to continued progress in rehabilitative care of persons with PD.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 70 years
* Willingness to spend 1-h in a scanner
* Able to walk with or without an assistive device 10 feet
* Best corrected/aided acuity better than 20/70 in the better eye
* Absence of dementia or vascular cognitive impairment
* Absence of primary memory deficits

Exclusion Criteria:

* Deep brain stimulator implants, Metallic implants, fragments, or pacemakers
* Montreal Cognitive Assessment (MocA) score < 24
* Pure-tone threshold sensitivity > 40 dB
* Peripheral neuropathy
* Untreated Major Depression
* History of stroke, or traumatic brain injury

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine E. Hackney, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Prime M, McKay JL, Bay AA, Hart AR, Kim C, Abraham A, Hackney ME. Differentiating Parkinson Disease Subtypes Using Clinical Balance Measures. J Neurol Phys Ther. 2020 Jan;44(1):34-41. doi: 10.1097/NPT.0000000000000297. PMID 31834219

RESULTS

PARTICIPANT FLOW:
Groups:
- Internally Guided Training (IG): Adapted tango dancing is a sophisticated, yet accessible system of tactile communication that conveys motor intentions and goals between a leader and follower. Those in IG training will choose direction, timing and amplitude of each successive step, and will communicate this information to their partner through moving their frame and center of mass.
  Adapted Tango Dancing: Composed of simple steps, tango involves frequent movement initiation and cessation, multi-directional perturbations and varied rhythms. Participants focus on trunk control and stepping strategies, coordination, somatosensory awareness, attention to partner, path of movement, and aesthetics. Sessions will begin with a typical dance class warm-up consisting of breathing, limbering and postural alignment to upbeat music. Novel step elements will be introduced every class period. Those with PD will partner with an individual without PD. After novel step introduction, the instructor will present rhythmic training, which is indispensable to partnered dancing. Participants will learn 'typical' rhythms from tango and Latin dances, based upon the system of quicks (Q) and slows (S), ubiquitously used in ballroom dance training to understand the temporal relationship of movement to music.
Period: Training
Arm/Group | Internally Guided Training (IG) | Externally Guided Training (EG) | Behavioral Control (BC)
Started | 34 | 31 | 22
Completed | 24 | 25 | 19
Not Completed | 10 | 6 | 3
Not completed — Lost to Follow-up | 10 | 6 | 3
Period: One Month Washout
Arm/Group | Internally Guided Training (IG) | Externally Guided Training (EG) | Behavioral Control (BC)
Started | 24 | 25 | 19
Completed | 24 | 24 | 18
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internally Guided Training (IG) | Externally Guided Training (EG) | Behavioral Control (BC) | Total
Number analyzed (Participants) | 34 | 31 | 22 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.0) | 68.6 (8.5) | 68.0 (9.5) | 69.36 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 6 | 33
  Male | 21 | 17 | 16 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 34 | 30 | 22 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 6 | 6 | 4 | 16
  White | 26 | 22 | 16 | 64
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Signal Change
Description: Percentage of baseline BOLD signal across activated brain regions. Activation values that remain significant after type-I error control in imaging software are averaged across brain regions, converted to Percent Signal Change, and presented as Mean (%) ± SD (%) across brain regions investigated.
Time Frame: 12 weeks
Population: The number of patients included in analyses is smaller than the total number of study participants due to study attrition and inability to tolerate the scanner.
Measure: Mean (Standard Deviation); unit: percentage of baseline BOLD signal
Arm/Group | Internal Guidance Training (IG) | Externally Guided Training (EG) | Behavioral Control (BC)
Number analyzed (Participants) | 19 | 19 | 17
percentage of baseline BOLD signal | 0 (0) | 23 (68) | 35 (44)

2. Primary Outcome: Connectivity Strength
Description: Changes in average connectivity strength across striatal-thalamo-cortical (STC) and cerebello-thalamo-cortical (CTC) circuits, as measured by average cross correlation coefficient between the seed regions of the circuits.
Time Frame: 12 weeks
Population: Sample size reflects study attrition and inability to tolerate fMRI scanning
Measure: Mean (Standard Deviation); unit: correlation coefficient
Groups:
- Behavioral Control: Dose-matched education courses
Arm/Group | Internal Guidance Training (IG) | Externally Guided Training (EG) | Behavioral Control
Number analyzed (Participants) | 20 | 21 | 17
correlation coefficient | -0.04 (0.51) | -0.03 (0.43) | 0.14 (0.34)

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time of study entry until the end of study participation, an average of 16 weeks.
Arm/Group | Internal Guidance Training (IG) | Externally Guided Training (EG) | Behavioral Control (BC)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/22
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT02457832/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT02457832/ICF_000.pdf